CLINICAL TRIAL: NCT04813146
Title: Role of Synchronized Lifestyle Modification Program on Diabetic Peripheral Neuropathy Patients Taking Oral Hypoglycemics and GLP-1 Analogues
Brief Title: Role of Synchronized Lifestyle Modification Program on Diabetic Neuropathy Taking Oral Hypoglycemics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRC/20/234 Rubab Rameez
Record Dates: First submitted 2021-02-02; First posted 2021-03-24 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Diabetic Neuropathies
Keywords: Synchronized Lifestyle Modification Program; Diabetic Neuropathy; Oral Hypoglycemic Agents
MeSH Terms: conditions — Diabetic Neuropathies | interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Synchronized Lifestyle Modification Program (SLP) (Experimental): Synchronized Lifestyle Modification Program ( Synchronization of dietary intake with the natural circadian rhythm of the body)
  Interventions: Other: SLP
- Synchronized Lifestyle Modification Program along with Physiotherapy (Experimental): Synchronized Lifestyle Modification Program along with Physiotherapy (Synchronization of dietary intake and Physiotherapy including aerobic, resistance, flexibility and balance exercises)
  Interventions: Other: SLP along with Physiotherapy
- Physiotherapy (Experimental): Physiotherapy (aerobics, resistance, flexibility and balance exercises)
  Interventions: Other: Physiotherapy
- Control Group (No Intervention): No Intervention will be given to this group ( conventional medicine will be given to these patient )

INTERVENTIONS:
Other: SLP — Synchronization of dietary intake with circadian rhythm of the body
  Arms: Synchronized Lifestyle Modification Program (SLP)
Other: SLP along with Physiotherapy — Synchronization of dietary intake along with Physiotherapy (aerobic, flexibility, resistance and balance exercises)
  Arms: Synchronized Lifestyle Modification Program along with Physiotherapy
Other: Physiotherapy — Physiotherapy given only (aerobic, flexibility, resistance and balance exercises)
  Arms: Physiotherapy

SUMMARY:
The aim of this study is to determine the combined effect of SLP along with Physiotherapy in improving Type 2 DPN patients taking OHAs and GLP-1 analogues.

DETAILED DESCRIPTION:
Diabetes mellitus (DM) is a chronic metabolic disease defined by persistently increased blood glucose levels with fasting blood glucose ≥ 126 mg/dl, random plasma glucose ≥ 200mg/dl and HbA1c ≥ 6.5%.

Diabetes has emerged as a great socioeconomic burden for the developing world. In 2017, globally, 451 million people were affected with diabetes. In Pakistan, the prevalence of type 2 diabetes is 16.98% which differs significantly with age, education, body mass index (BMI), obesity, family history and blood pressure. DM is classified into type 1 diabetes (T1D) and type 2 diabetes (T2D). T1D occurs due to an autoimmune pancreatic beta cell destruction with consequent insulin deficiency whereas T2D occurs due to predominantly insulin resistance with relative insulin deficiency or defective secretion. T2D cause serious and chronic microvascular and macrovascular complications. One of the most prevalent microvascular complication is diabetic peripheral neuropathy (DPN). DPN is defined as distal, symmetric sensorimotor polyneuropathy as a result of hyperglycemia and microangiopathy. It is a demyelinating disease of peripheral nerve fibers that manifests as parasthesias, impairment of sensations of vibration, proprioception, touch, pressure, pain and temperature.

Risk factors of DPN are age, duration of diabetes, HbA1c >7.0%, increased BMI, hyperlipidemia and hyperglycemia. Treatment of T2D is targeted towards good glycemic control that includes life style modifications i.e. diet and exercise, oral hypoglycemic agents (OHAs) and subcutaneous insulin administration. In life style modification, variety of exercises are recommended that help to slow the progression of peripheral neuropathy.These include; aerobic training, weight-bearing, static and dynamic balance training and strength training exercises which improve the gait speed, stride length and nerve conduction velocities (NCVs) of sensory and motor nerves while flexibility exercises improve the range-of-motion in ankle, hip and shoulder joints and keep them flexible. Importance of dietary modification is enhanced if it is synchronized with the circadian rhythm of the body. Therefore, Synchronized Lifestyle Modification Program (SLP) is a personalized, homeostasis restoring, liver centric lifestyle modification program that works through the correction of body clock rhythm. Lifestyle medicine is defined as the discipline of studying how daily habits and practices impact both on the prevention and treatment of disease. Its key aspects are: regular physical activity, proper nutrition, weight management, avoiding tobacco and a sound mental health. Lifestyle modification in diabetics is believed to enhance the function of pancreatic islet cells and induce glucose-stimulated insulin release.Regarding pharmacological treatment, following OHAs are used which are; biguanides, insulin secretagogues, alpha-glucosidase inhibitors, thiazolidinediones, dipeptidyl peptidase-4 (DPP4) inhibitors and sodium glucose co-transporter-2 inhibitors. Now a days, an injectable agent i.e. Glucagon like peptide-1(GLP-1) receptor agonist is used with OHAs and is effective in decreasing blood glucose levels with a low risk of hypoglycemia in elderly patients.

Limited data is available which supports the combined effect of Synchronized Lifestyle modification Program (SLP) and Physiotherapy in the progression of DPN in T2D patients taking OHAs and GLP-1.

ELIGIBILITY:
Inclusion Criteria:

* Gender includes both male and female
* Patients between age group 40-75 years
* Clinically diagnosed patients of Type 2 diabetes on OHAs and GLP-1 analogues
* Diabetic patients with symptomatic peripheral neuropathy (Severity of DPN is associated with a physical examination score > 2.5 by using Michigan Neuropathy Screening Instrument (MNSI) with grades mild, moderate and severe)

Exclusion Criteria:

* Type 1 diabetic patients
* Age < 40 years and > 75 years
* Patients with any other co-morbidities (Heart, liver and kidney diseases)
* Patients with neuropathies due to any other disease
* Orthopaedic and surgical procedure of lower limbs
* Patients with foot ulcers
* Peripheral vascular diseases
* Patients receiving any structured supervised physiotherapy
* Pregnant females

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2021-02-05 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
Life style pattern assessment | 12 weeks
  Changes from baseline, assessed through a self-structured questionnaire consisting of open-ended questions to assess the timing and type of food taken in meals, daily water intake and sleeping habits. Total 10 questions are included.
Calculation of Body Mass Index | 12 weeks
  Changes from baseline calculated by measuring height in meters through a metal measuring tape and weight in kilograms through portable manual weighing scale. BMI with minimum value of 18.5 kilogram/ meters square (kg/m2) and maximum value of 24.9 kilogram /meters square (kg/m2). Below 18.5 kilograms/meters square (kg/m2) is considered as underweight and above 24.9 kilogram/meters square (kg/m2) is considered as obese.
Measurement of Systolic Blood pressure | 12 weeks
  Changes from baseline are assessed by using Mercury Sphygmomanometer with minimum value of 110 millimeter of mercury (mmHg) and the maximum value of 130 millimeter of mercury (mmHg). Below 110 millimeter of mercury (mmHg) is considered as low systolic blood pressure and above 130 millimeter of mercury (mmHg) is considered as high systolic blood pressure.
Measurement of Diastolic Blood pressure | 12 weeks
  Changes from baseline are assessed by using Mercury Sphygmomanometer with minimum value of 60 millimeter of mercury (mmHg) and the maximum value of 90 millimeter of mercury (mmHg). Below 60 millimeter of mercury (mmHg) is considered as low diastolic blood pressure and a value above 90 millimeter of mercury (mmHg) is considered as high diastolic blood pressure.
Michigan Neuropathy Screening Instrument | 12 weeks
  Changes from baseline is assessed. Subjective assessment is done by a questionnaire that is self-administered by the participants. Responses of "yes" are given to questions 1-3, 5-6, 8-9, 11-12, 14-15 and each of them counted as one point. A "no" response is given on questions 7 and 13 and are counted as 1 point. A score of more than or equal to 7 in the history questionnaire is considered abnormal. Lower extremity examination includes inspection and assessment of vibratory sensation and ankle reflexes which is considered as abnormal at a score of more than or equal to 2.5.
Peak latency of Sensory Nerves (Sural and Peroneal) | 12 weeks
  Changes from baseline is assessed through nerve conduction studies. Value of 4.2 millisecond (ms) of sural nerve and 6.1 millisecond (ms) for peroneal nerve is considered normal. Values below 4.2 millisecond (ms) and 6.1 millisecond (ms) are considered abnormal.
Amplitude of Sensory Nerves (Sural and Peroneal) | 12 weeks
  Changes from baseline are assessed through nerve conduction studies with a value of 6 microvolt (µV) for sural nerve and 2 microvolt (µV) for peroneal are considered normal. Values below 6 microvolt (µV) and 2 microvolt (µV) are considered abnormal.
Velocity of Sensory Nerves | 12 weeks
  Changes from baseline are assessed through nerve conduction studies with value of 41 meters/second (m/sec) is considered normal. Value below 41meters/second (m/sec) is considered abnormal.
Onset Latency of Motor Nerves (Peroneal and Tibial) | 12 weeks
  Changes from baseline are assessed through nerve conduction studies with value of 6.1 millisecond (ms) for both are considered normal. Value below 6.1 millisecond (ms) is considered abnormal.
Amplitude of Motor Nerves (Peroneal and Tibial) | 12 weeks
  Changes from baseline are assessed through nerve conduction studies with values of 2 millivolt (mV) and 3 millivolt (mV) are considered normal. Values below 2 millivolt (mV) and 3 millivolt (mV) are considered abnormal.
Velocity of Motor Nerves (Peroneal and Tibial) | 12 weeks
  Changes from baseline are assessed through nerve conduction studies with values of 41 meters/second (m/sec) is considered normal for both nerves. Value less than 41 meters/second (m/sec) is considered abnormal.
Assessment of Balance by Berg Balance Scale | 12 weeks
  Changes from baseline are assessed with Low Fall Risk 41-56, Medium Fall Risk 21-40, High Fall Risk 0-20.
Serum Fasting Blood Glucose | 12 weeks
  Changes from baseline are measured by Glucose oxidase enzyme based method in milligram/deciliter (mg/dL) using Glucometer with minimum value of 72 milligram/deciliter (mg/dL) and maximum value of 99 milligram/deciliter (mg/dL). Value below 72 milligram/deciliter (mg/dL) is considered hypoglycemic and above 99 milligram/deciliter (mg/dL) is hyperglycemic.
Serum Total Cholesterol | 12 weeks
  Changes from baseline are measured by Cholesterol oxidase enzyme based method with minimum value of 125 milligram/deciliter (mg/dL) and maximum value of 200 milligram/deciliter (mg/dL).
Serum Triglycerides | 12 weeks
  Changes from baseline are measured by Glycerol phosphate enzyme based method with minimum value of less than150 milligram/deciliter (mg/dL) and maximum value of199 milligram/deciliter (mg/dL).
Serum High Density Lipoproteins (HDL) | 12 weeks
  Changes from baseline are measured by Direct enzymatic immune-inhibition with minimum value of 40 milligram/deciliter (mg/dL) and maximum value of greater than 40 milligram/deciliter (mg/dL).
Serum Low Density Lipoproteins | 12 weeks
  Changes from baseline are measured by Friedewald calculation with minimum value of 100 milligram/deciliter (mg/dL) and maximum value of 129 milligram/deciliter (mg/dL).
Serum HbA1c concentration | 12 weeks
  Changes from baseline are measured by Ion exchange chromatography with minimum value of 4 % and maximum value of 5.9 %. Normal range for the HbA1c level is between 4% and 5.6%. Levels between 5.7% and 6.4% is the pre-diabetic range. Levels of 6.5% or higher is diabetic range.

CONTACTS AND LOCATIONS:
Overall Officials: Shazia Ali, PhD, Principal Investigator — Riphah International University
Locations (1):
- Pakistan Railway Hospital, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Khawandanah J. Double or hybrid diabetes: A systematic review on disease prevalence, characteristics and risk factors. Nutr Diabetes. 2019 Nov 4;9(1):33. doi: 10.1038/s41387-019-0101-1. PMID 31685799
- [Background] Aamir AH, Ul-Haq Z, Mahar SA, Qureshi FM, Ahmad I, Jawa A, Sheikh A, Raza A, Fazid S, Jadoon Z, Ishtiaq O, Safdar N, Afridi H, Heald AH. Diabetes Prevalence Survey of Pakistan (DPS-PAK): prevalence of type 2 diabetes mellitus and prediabetes using HbA1c: a population-based survey from Pakistan. BMJ Open. 2019 Feb 21;9(2):e025300. doi: 10.1136/bmjopen-2018-025300. PMID 30796126
- [Background] Diabetes Canada Clinical Practice Guidelines Expert Committee; Punthakee Z, Goldenberg R, Katz P. Definition, Classification and Diagnosis of Diabetes, Prediabetes and Metabolic Syndrome. Can J Diabetes. 2018 Apr;42 Suppl 1:S10-S15. doi: 10.1016/j.jcjd.2017.10.003. No abstract available. PMID 29650080
- [Background] Iqbal Z, Azmi S, Yadav R, Ferdousi M, Kumar M, Cuthbertson DJ, Lim J, Malik RA, Alam U. Diabetic Peripheral Neuropathy: Epidemiology, Diagnosis, and Pharmacotherapy. Clin Ther. 2018 Jun;40(6):828-849. doi: 10.1016/j.clinthera.2018.04.001. Epub 2018 Apr 30. PMID 29709457
- [Background] Cancelliere P. A Review of the Pathophysiology and Clinical Sequelae of Diabetic Polyneuropathy in the Feet. J Diabetes, Metab Disord Control. 2016;3(2):21-4.
- [Background] Liu X, Xu Y, An M, Zeng Q. The risk factors for diabetic peripheral neuropathy: A meta-analysis. PLoS One. 2019 Feb 20;14(2):e0212574. doi: 10.1371/journal.pone.0212574. eCollection 2019. PMID 30785930
- [Background] Qaseem A, Barry MJ, Humphrey LL, Forciea MA; Clinical Guidelines Committee of the American College of Physicians; Fitterman N, Horwitch C, Kansagara D, McLean RM, Wilt TJ. Oral Pharmacologic Treatment of Type 2 Diabetes Mellitus: A Clinical Practice Guideline Update From the American College of Physicians. Ann Intern Med. 2017 Feb 21;166(4):279-290. doi: 10.7326/M16-1860. Epub 2017 Jan 3. PMID 28055075
- [Background] Gholami F, Nikookheslat S, Salekzamani Y, Boule N, Jafari A. Effect of aerobic training on nerve conduction in men with type 2 diabetes and peripheral neuropathy: A randomized controlled trial. Neurophysiol Clin. 2018 Sep;48(4):195-202. doi: 10.1016/j.neucli.2018.03.001. Epub 2018 Mar 30. PMID 29606547
- [Background] Majeedkutty NA, Jabbar MA, Sreenivasulu S. Physical therapy for diabetic peripheral neuropathy: A narrative review. Disabil CBR Incl Dev. 2019;30(1):112-25.
- [Background] Bae SA, Fang MZ, Rustgi V, Zarbl H, Androulakis IP. At the Interface of Lifestyle, Behavior, and Circadian Rhythms: Metabolic Implications. Front Nutr. 2019 Aug 28;6:132. doi: 10.3389/fnut.2019.00132. eCollection 2019. PMID 31555652
- [Background] Parr EB, Heilbronn LK, Hawley JA. A Time to Eat and a Time to Exercise. Exerc Sport Sci Rev. 2020 Jan;48(1):4-10. doi: 10.1249/JES.0000000000000207. PMID 31688298
- [Background] Rippe JM. Lifestyle Medicine: The Health Promoting Power of Daily Habits and Practices. Am J Lifestyle Med. 2018 Jul 20;12(6):499-512. doi: 10.1177/1559827618785554. eCollection 2018 Nov-Dec. PMID 30783405
- [Background] Marin-Penalver JJ, Martin-Timon I, Sevillano-Collantes C, Del Canizo-Gomez FJ. Update on the treatment of type 2 diabetes mellitus. World J Diabetes. 2016 Sep 15;7(17):354-95. doi: 10.4239/wjd.v7.i17.354. PMID 27660695